CLINICAL TRIAL: NCT04118179
Title: Development of a New Strategy to Predict Early Sepsis
Brief Title: New Strategy to Predict Early Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bob Hancock, Canada Research Chair and Professor, Department of Microbiology and Immunology, University of British Columbia
Other Study IDs: H17-01208
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA samples obtained from whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspected Sepsis Group: Participants suspected of potential to develop sepsis recruited at the emergency department.
  Interventions: Other: Blood sample collection
- Surgical Group: Participants undergoing non-emergency scheduled surgery, including ear/nose and throat cases, orthopaedic surgery of the major joints including hip, knee, ankle, shoulder, and wrist.
  Interventions: Other: Blood sample collection
- Healthy Group: Healthy participants
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — A blood sample (1 tube) will be collected for the analysis of the CR signature.

SUMMARY:
This is an observational prospective multicentre study on patients attending the emergency department and suspected to have sepsis. Blood markers characteristic of a Cellular Reprogramming (CR) signature and predicting severe sepsis and organ failure will be measured and validated.

DETAILED DESCRIPTION:
Sepsis is a life-threatening medical condition caused by an infection and the complex and dysfunctional way by which the human body attempts to deal with it. It can affect people of all ages, causing 18-30 million cases and 5-8 million deaths annually worldwide. However, early diagnosis of sepsis is challenging due to the diversity and overlap of symptoms with other disorders and the lack of an early and accurate diagnostic method. Hancock and colleagues defined a gene expression signature characteristic of biological changes occurring during sepsis, known as cellular reprogramming (CR) and reflecting a type of immune amnesia (inability to respond to bacterial signals). This signature was shown to predict the development of sepsis and organ failure at first clinical presentation in the emergency room, by examining patient blood samples taken during an initial pilot single-center study.

This project will validate and refine the CR signature and demonstrate reproducibility, specificity, and sensitivity in a larger multi-center study to enable a new strategy to predict Sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Presenting to the Emergency Department
* Attending physician suspects possible sepsis based on at least 2 sign of Systemic inflammatory response syndrome (SIRS) criteria and suspicion of infection

Exclusion Criteria:

* Patient is terminal (death anticipated in 12 hours)
* Informed consent unobtainable if the subject survives to hospital discharge.
* Subjects who are unable to provide blood as a standard of care.
* Blood sample could not be taken within 24 hours of a physician's first contact with the patient.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suspected of sepsis will be recruited at the emergency department of participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Severity of illness | 24 hours
  Measured by serial Sequential Organ Failure Assessment (SOFA) score monitoring

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) Score monitoring | 72 hours
  The organs scored are respiratory, cardiovascular, neurologic, hematologic, renal, and liver. Each organ is scored as 0 (best) to 4 (worse) and the total score is the sum of each component.
Mortality | 28 days
  28-day survival rate after admission to hospital
ICU length of stay | 28 days
  Length of stay in the Intensive Care Unit
Quick Sequential Organ Failure Assessment (SOFA) Score greater than 2 | 6 hours
  Measured by serial Sequential Organ Failure Assessment (SOFA) score monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Hancock, PhD, Principal Investigator — University of British Columbia
Locations (5):
- University of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States
- Westmead Hospital, Sydney, Australia
- Vancouver General Hospital, Vancouver, Canada
- Hospital Universitario Moncaleano Perdomo, Neiva, Colombia
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The RNA-Seq data will be uploaded to Geo database when the study is complete or upon publication and will be freely available to researchers.

REFERENCES:
- [Background] Pena OM, Hancock DG, Lyle NH, Linder A, Russell JA, Xia J, Fjell CD, Boyd JH, Hancock RE. An Endotoxin Tolerance Signature Predicts Sepsis and Organ Dysfunction at Initial Clinical Presentation. EBioMedicine. 2014 Nov 1;1(1):64-71. doi: 10.1016/j.ebiom.2014.10.003. PMID 25685830